CLINICAL TRIAL: NCT06021132
Title: Characterisation of Low Frequency Hearing and Vestibular Function in Patients Undergoing Cochlear Implantation
Status: Active, not recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jonas Bruun Kjærsgaard, MD, Aalborg University Hospital
Other Study IDs: RN-86132
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: Cochlear implant; Residual hearing; Hearing preservation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: cochlear implant — Insertion of a electrode into the cochlear with the aim of providing deaf and severe hearing handicapped with the ability to hear speech.

SUMMARY:
The study will follow a cohort of CI-candidates becoming CI-user, till two years postoperative. A through-out assessment of both their audiological and vestibular status will be carried out at multiple fixed timepoints over 2 years, evaluating both subjective (patients reported) and objective outcomes over time. For the audiological part of the study both pure-tone and speech audiometry results will be held against the patient perceived benefit of the treatment as assessed by the questionnaires NCIQ and SSQ-12. The vestibular part of the study will evaluate the function of the SCCs and the sacculus. This is will be put in concert with functional tests of the vestibular system, and the patient perceived outcome measure DHI. Correlations between vestibular and audiological performances will be examined. A collection of specific hypotheses will be tested by predefined statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Adults (At or above 18 years of age and capable of giving an informed consent)
* Cochlear implant candidacy
* Profound bilateral post-lingual hearing loss
* Proficiency in Danish
* Expected ability to participate on both all pre- and postoperative examinations
* No previous CI experiences

Exclusion Criteria:

* Later abandonment of CI candidacy
* Blindness or visual handicap compromising eye movement evaluation
* Distinct neck mobility handicap hindering either vHIT- or cVEMP examination
* Patient reluctance, such as consistent no-show or cancellations of appointments
* CI-surgery before preoperative evaluation could be obtained
* Simultaneous bilateral cochlea implantation.
* Sequential CI within the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CI-candidates are to be included from our tertiary referral centre at the Audiological Department at Aalborg University Hospital, Aalborg, Denmark.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Anticipated increase in speech audiometric performances | +24 months from last inclusion. Expected to be complete in juli 2025.
  The preoperative status will be held against their performance at 6, 12 and 24 months. Yet the performance at 6 months will also be held against status at 24 months
Anticipated increase in patient reported outcome measures | +24 months from last inclusion. Expected to be complete in juli 2025.
  The preoperative status will be held against their performance at 6, 12 and 24 months. Yet the performance at 6 months will also be held against status at 24 months
Test-retest assessment of vestibular screening battery | Conducted before cochlear implantation in all patients.
  Double examination using commercial video head impulse test system and cervical vestibular evoked myogenic potentials.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas B Kjlærsgaard, MD, Principal Investigator — ENT department, Aalborg University Hospital; Michael L Gaihede, PhD, MD, Study Director — ENT department, Aalborg University Hospital
Locations (1):
- Balance & Dizziness Centre, Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Full plan of analysis and raw data will be presented given there is still anonymity for the participants.